CLINICAL TRIAL: NCT06820138
Title: Low Intensity Focused Ultrasound for Posttraumatic Stress Disorder
Brief Title: Focused Ultrasound for PTSD in Veterans
Acronym: PTSD FUS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N5299-R
Record Dates: First submitted 2025-01-27; First posted 2025-02-11 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Low intensity focused ultrasound
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Double-blind delivery of low intensity focused ultrasound (i.e., active low intensity focused ultrasound versus a sham (placebo) administration of low intensity focused ultrasound). Sessions are approximately three times a week for four weeks.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Identical active and sham transducer pads are used; these are pads used to couple the ultrasound device to the participant. Sham pads have material that does not permit ultrasound energy to pass through
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Verum low intensity focused ultrasound (Active Comparator): Verum (active) low intensity focused ultrasound, applied up to three times per week.
  Interventions: Device: Brainsonix Ultrasound Device
- Sham low intensity focused ultrasound (Sham Comparator): Sham (inactive) low intensity focused ultrasound, applied up to three times per week.
  Interventions: Device: Brainsonix Ultrasound Device

INTERVENTIONS:
Device: Brainsonix Ultrasound Device — This device delivers low intensity focused ultrasound and delivers either active or sham sonication depending upon the transducer pad used.
  Other Names: Brainsonix Pulsar

SUMMARY:
The goal of this study is to develop a new, non-invasive brain stimulation modality called low intensity focused ultrasound (FUS) as a psychiatric rehabilitation treatment for posttraumatic stress disorder (PTSD). FUS delivers energy comparable to that involved in diagnostic ultrasound but in a millimeter-sized envelope. Unlike currently available methods, the maximal FUS energy is delivered at a distance from a transducer on the scalp. Therefore, its promise is that it can deliver focal and reversible modulation to deeper brain regions involved in PTSD. The investigator team has previously conducted first-in-human research in FUS, and this study builds upon that work to conduct a phase II, dose-finding study. This study will pursue two Aims; the first is whether FUS to the amygdala can improve symptoms, and the second will evaluate whether FUS improves function by reduced disability, over a 1-month period. Short and longer-term effects of FUS will be measured and all FUS parameters are within FDA-defined safety thresholds for diagnostic ultrasound.

DETAILED DESCRIPTION:
PTSD is highly prevalent in Veterans and is associated with significant psychiatric and medical comorbidity and healthcare utilization. Most importantly, PTSD prevents Veterans from reintegrating into society and is associated with significant disability and psychosocial dysfunction. Despite its prevalence and devastating impact, even the most efficacious treatments have modest success in improving either symptoms or functioning in Veterans with PTSD. One reason for this limited efficacy is the inability for current treatments to directly target and engage deep brain regions which are directly involved in PTSD psychopathology. However, recent advances in the areas of neuroscience, psychiatry and technology allow, for the first time, development of new technologies that can non-invasively and reversibly modulate deep brain structures through the use of low intensity focused ultrasound (FUS). This application is targeting the amygdala, which is a core region involved in PTSD and many other psychiatric disorders.

To date, cleared uses of focused ultrasound are high-intensity sonication to irreversibly ablate tissue, therapeutically for movement disorders and cancer-related pain. Effects are highly focal (i.e., millimeter-scale), and occur without adjacent tissue damage. In contrast, FUS as it is proposed here uses acoustic energy at the same precision but within safety limits for diagnostic ultrasound. Although therapeutic use of FUS remains largely unexplored, several groups demonstrated that FUS can safely modulates neural activity in mice, rabbit, swine, and non-human primates. Even more recent data indicates FUS can safely modulate human cortical activity, including that of somatosensory and motor cortex as well as the thalamus in healthy individuals.

Our group has been leading the effort to evaluate the use of FUS, by delivering a single dose of FUS inside the bore of an MRI scanner to a group of depressed Veterans. However, FUS has not yet been developed for PTSD, and before rigorous clinical trials of FUS for PTSD can be initiated, several key questions remain and are the focus of this study.

Using a phase II-style proof of concept/dose-finding study, investigators will characterize the effects of sham-controlled FUS administrations. Veterans with chronic PTSD first receive an MRI scan to facilitate high-precision targeting using out-of-scanner stereotactic neuronavigation. After targeting, Veterans are randomized to receive sham FUS, or one, two, or three FUS administrations per week over a month, and then Veterans will be followed for up to three months to evaluate longer-term effects. Neuroimaging MRI will be obtained prior to and following completion of FUS to explore neural effects. Thus, this study will evaluate the short-term durability of any effects on symptoms and function, and the design will provide important insight into the potential use for repeated administrations over time. The significance of this project lies in the potential to develop non-invasive deep brain stimulation for PTSD, with lessons learned that will be applicable for broader implementation; this goal can be realized through this careful and programmatic phase II study.

ELIGIBILITY:
Inclusion Criteria:

-Veterans ages 22-70 (inclusive) who meet DSM-5 criteria for chronic PTSD using the Clinician Administered PTSD Scale for DSM-5 (CAPS-5) and currently symptomatic. If applicable, Veterans will be required to be on stable psychiatric treatment(s) prior to baseline assessments

Exclusion Criteria:

* contraindications to focused ultrasound and/or neuroimaging:

  * i) history of seizure disorder or serious neurologic illness including dementia or serious cognitive impairment,
  * ii) structural or neurologic abnormalities present or in close proximity to sonication site ,
  * iii) prior brain surgery,
  * iv) pacemaker or implanted central nervous system device,
  * v) greater than mild traumatic brain injury, or any head injury within sixty days of ultrasound,
  * vi) greater than moderate alcohol or substance use disorders or active use or withdrawal from alcohol or substances,
  * vii) metal in the head,
  * viii) physical impediment likely to interfere with assessments, or
  * ix) unable to follow protocols.
  * x) Veterans with significant white matter findings or those with findings in the beam of the ultrasound may also be excluded at discretion of study staff.
* Veterans with acute suicidality are also excluded.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-08-03 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-03-29 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist for DSM5 | Up to 3 months
  The PTSD Checklist for Diagnostic and Statistical Manual-5 (PCL-5) is a gold standard self reported scale of PTSD symptoms. Scores range from 0-80, where higher scores indicate greater symptom severity. The Week 5 visit value is the primary outcome measure of the study.

SECONDARY OUTCOMES:
Sheehan Disability Scale | Up to 3 months
  The Sheehan Disability Scale (SDS) is a self report tool used to assess functional impairment in work, social and family life. Scores range from 0-30, where higher scores indicate greater impairment.
Social and Occupational Function Scale | Up to 3 months
  The Social and Occupational Function Scale (SOFAS) assesses social and occupational function, and is scored from 0-100, where higher scores indicate superior (better) social and occupational function.
Inventory of Depressive Symptoms Self Report | Up to 3 months
  The Inventory of Depressive Symptoms, Self-Report (IDSSR) is a rating scale that measures self-reported depressive symptoms. Scores range from 0-84, where higher scores indicate more severe depressive symptom severity.
Clinician Administered PTSD Scale | Up to 3 months
  The Clinician Administered Posttraumatic Stress Disorder Scale for Diagnostic and Statistical Manual-5 (CAPS-5) is structured clinical interview for posttraumatic stress disorder symptoms. Scores range from 0-80, where higher symptoms indicate more severe symptom severity.
Clinician Global Impression | Up to 3 months
  The Clinician Global Impression scale assesses a clinician's general impression of severity. Scores typically range from 1 (not at all ill) to 7 (very ill); Improvement scores range from 1 (very much improved) to 7 (very much worse).

OTHER OUTCOMES:
Visual Analog Scale | Three times per week for up to five weeks
  The visual analog scale assesses global symptom burden and is assessed immediately after ultrasound administration. Scores are rated on a visual scale from 0 to 100 where 100 is the maximum global burden.
Arterial Spin Labeling/fMRI | Five weeks
  Functional magnetic resonance imaging measures are assessed prior to and following all focused ultrasound procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Noah S. Philip, MD, Principal Investigator — Providence VA Medical Center, Providence, RI
Locations (1):
- Providence VA Medical Center, Providence, RI, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No